CLINICAL TRIAL: NCT01863160
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Dose-escalating Study to Assess Safety, Tolerability and Pharmacokinetics of 0.1% and 1.0% ZEP-3 Cream, Administered Topically in Healthy Volunteers.
Brief Title: Safety and Tolerability Study of ZEP-3 Cream (0.1% and 1.0%), Administered Topically In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shulov Innovate for Science Ltd. 2012 (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: ZEP - 001 - IL
Record Dates: First submitted 2013-05-13; First posted 2013-05-27 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetic profile; ZEP-3 Cream (0.1% and 1.0%); administered topically

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.1% ZEP-3 cream (Other): 250 mg of ZEP-3 Cream 0.1% is applied on the right ventral forearm and 250 mg placebo is applied on the left ventral forearm 4 times daily
  Interventions: Drug: 0.1% ZEP-3 cream
- placebo (Other): 250 mg of ZEP-3 Cream 1.0% is applied on the right ventral forearm and 250 mg placebo is applied on the left ventral forearm 4 times daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 0.1% ZEP-3 cream — Topical application of 250mg ZEP-3 cream (0.1%) vs. placebo 4 times daily The IP is applied to "in advanced" demarcated sites in a dose escalating mode to 3 different treatment area sizes: small area of 2x1 cm (2 cm2), medium area of 2x5 cm (10 cm2), and large area of 4x5 cm (20 cm2).
  The IP ZEP-3 cream will be applied on both ventral forearms (one application site per forearm) in a non-occlusive mode, spread and rubbed over the demarcated area.
  * Right arm, single treatment area - ZEP-3 (0.1%)
  * Left arm, single treatment area - Placebo cream
  Other Names: novel synthetic peptide
  Arms: 0.1% ZEP-3 cream
Drug: placebo — Topical application of 250mg ZEP-3 cream (1.0%) vs. placebo 4 times daily The IP is applied to "in advanced" demarcated sites in a dose escalating mode to 3 different treatment area sizes: small area of 2x1 cm (2 cm2), medium area of 2x5 cm (10 cm2), and large area of 4x5 cm (20 cm2).
  The IP ZEP-3 cream will be applied on both ventral forearms (one application site per forearm) in a non-occlusive mode, spread and rubbed over the demarcated area.
  Right arm, single treatment area - ZEP-3 (1.0%)
  Left arm, single treatment area - Placebo cream
  Other Names: novel synthetic peptide
  Arms: placebo

SUMMARY:
It is a phase I randomized, double blind, placebo-controlled, dose-escalating study to assess safety, tolerability and pharmacokinetics (PK) data of 0.1% and 1.0% ZEP-3 cream, administered topically up to 5 consecutive treatment days in healthy volunteers.

This is a single center trial. It is anticipated that the study will be conducted at the Department of Dermatology, at the Sheba Medical Center, Ramat Gan, Israel.

The screening/enrollment visit includes a PK study for 24h following a single IP topical application. After a 24h washout time break, the subject will enter the treatment period for 5 consecutive treatment days followed by a follow up visit 1 and 5 days after end of treatment.

DETAILED DESCRIPTION:
The primary endpoints of this study are:

* Safety evaluation - To demonstrate ZEP-3 cream safety in terms of skin irritation score.
* Safety evaluation - To demonstrate ZEP-3 cream safety in terms of type and severity of reported adverse events.
* Tolerability evaluation - To demonstrate ZEP-3 cream tolerability in terms of treatment compliance by the treated volunteers.

The secondary endpoints of this study are:

* Systemic absorption PK profile.
* Dermal absorption PK profile (Optional).

Subject safety will be assessed following treatment by ZEP-3 cream, using measurements of the following variables:

* Dermal reaction parameters
* Physical examination
* Vital Signs (HR, BP, RR, Body temperature)
* 12 lead ECG data
* Laboratory tests (CBC, blood chemistry, coagulation functions, urinalysis)
* Adverse events recording
* Change in concomitant medications

ELIGIBILITY:
Inclusion Criteria:

1. Subject must voluntarily sign and date the written Informed Consent prior to any study specific procedures
2. Subject, either men or women is between 18 and 50 years of age.
3. Subject, Body mass index (BMI) is within the normal to overweight range (See appendix 2)
4. Subject must have healthy skin on which reddening can be easily recognized in the area where they will place the test article
5. Subject must be free from a condition/disease that the investigator feels interferes with the interpretation of the study results.
6. Subject is willing to participate in the study and adhere to the study protocol
7. Females of childbearing potential should either be surgically sterile, or should use a highly effective medically accepted contraceptive regimen.

Exclusion Criteria:

1. Subject has hyper- or hypo-pigmentation, or tattoos in the area where they will place the test fields
2. Dark skinned persons whose skin color prevents ready assessment of skin reactions
3. Subject with history of skin disorders or any active skin condition involving the test fields including but not limited to bacterial, viral, or fungal skin infections, acne, rosacea
4. UV therapy or significant UV exposure in the four weeks before treatment application
5. Subject with renal failure (Cr > 2 mg/dl) or Subject with impaired hepatic function (ALT, AST 2-fold higher than normal upper limit value).
6. Cardiac disease, including recent myocardial infarction, any degree of heart block or other cardiac arrhythmias and valvular heart disease
7. Subject suffers from an autoimmune disease (Diabetes, Lupus. Chron ect.)
8. History of malignancy
9. Sever illness or surgery within the previous 3 months (except for minor cosmetic or dental procedures)
10. Treatment with any investigational agent in another clinical trial within 1 month prior to start of this study.
11. Female subject who is pregnant , lactating, or with a positive pregnancy test
12. History of drug or alcohol abuse (as defined by the Investigator)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Topical skin safety evaluation | Change in skin clinical presentation up to 5 consecutive treatment days
  Skin irritation

SECONDARY OUTCOMES:
Systemic absorption | During 24 hours following initial application
  PK profile

CONTACTS AND LOCATIONS:
Overall Officials: Aviv Barzily, PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel